CLINICAL TRIAL: NCT03410303
Title: Evaluation of Intraoperative Ultrasound for the Positioning of Prostheses in Laparoscopic Surgery of Genital Prolapse
Brief Title: Per-operative Ultrasonographic Assessement of the Placement of the Mesh in Laparoscopic Sacral Colpo/Hysteropexy
Acronym: SONOMESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K160801J
Record Dates: First submitted 2017-12-20; First posted 2018-01-25 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: LAPAROSCOPY; Sacrum; Anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative ultrasound (Other): An ultrasound of the position of the prosthesis during surgery, under general anesthesia, is performed. A follow-up visit will be carried out 2 months (± 1 month) after the surgery as part of the usual care. An ultrasound of the position of the prosthesis is performed without anesthesia, either as part of the treatment or as part of the research. This measurement is performed without the intraoperative measurement by an independent sonographer.
  Interventions: Diagnostic Test: Intraoperative ultrasound and 2 months post-operative ultrasound ( ± 1 month)

INTERVENTIONS:
Diagnostic Test: Intraoperative ultrasound and 2 months post-operative ultrasound ( ± 1 month) — An ultrasound of the position of the prosthesis during surgery, under general anesthesia, is performed. A follow-up visit will be carried out 2 months (± 1 month) after the surgery as part of the usual care. An ultrasound of the position of the prosthesis is performed without anesthesia, either as part of the treatment or as part of the research. This measurement is performed without the intraoperative measurement by an independent sonographer.

SUMMARY:
This study is conducted in order to determinate the faisability of an intraoperative ultrasound to mesure the positioning of prostheses during laparoscopic promontofixation.

DETAILED DESCRIPTION:
Genital prolapse is a very common functional pathology that affects 30% of women. The functional impact of prolapse is highly variable and may lead patients to consider surgery. Surgery for laparoscopic genital prolapse (laparoscopy) is a common practice. The placement of prostheses on the anterior and posterior walls of the vagina is sort of "estimated", performed without any quality control . This technique is associated with a high rate of patient satisfaction (90% satisfaction), but a risk of anatomical recurrence in 20-30% of cases and a risk of reoperation for relapse in 3% of cases. It is likely that the lower the intervesico-vaginal prosthesis, the lower the risk of cystocele relapse is important.The postoperative ultrasound visualization of prostheses placed in promontofixation is possible: they appear hyperechoic. In particular, in anterior, where a prosthesis is placed between the vagina and the bladder, it is possible to verify that this prosthesis supports the entire bladder base.Thus, it may be possible to check the correct position of the prostheses intraoperatively. If studies were conducted postoperatively, to the best of our knowledge, no study has been conducted on the value of an intraoperative ultrasound control.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (>18 years-old)
* patient who undergo laparoscopic sacral copopexy/hysteropexy
* Affiliation to a public health insurance system
* Written and informed consent given by the patient

Exclusion Criteria:

* Pregnancy, breast-feading
* woan involved in an interventional research
* Patient under tutorship or curatorship
* Pregnancy and breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Measure the distance (in mm) between the most distal part of the anterior prosthesis and the bladder neck. | at two months (± 1 month) of follow-up
  Comparaison of intraoperative measurement to postoperative measurement

SECONDARY OUTCOMES:
Stage of prolapse | until 2 months post-operative
  Evaluate the stage of prolapse on clinical examination according to the International Continence Society (ICS) of Pelvic Organ Prolapse Quantification System (POP-Q) classification (points Ba, Bp, C, D)
Evaluate the symptoms with the PFDI-20 questionnaire | during 2 months post-operative
  The Pelvic Floor Disorders Inventory (PFDI-20) score : This is a questionnaire so that patients can answer questions about certain symptoms: intestines, bladder or pelvic
Evaluate patient satisfaction with the PGI-I questionnaire (1-7) | until 2 months post-operative
  The Patient Global Impression of Improvement (PGI-I) : The patient should check the box corresponding to the current state of her uro-gynecological problems compared to what they were before treatment
Evaluate the symptoms with the PFIQ-7 questionnaire | during 2 months post-operative
  The Pelvic Floor Impact Questionnaire (PFIQ-7) : describe how much les activities, relationships, or feelings have been affected by symptoms bladder, bowel, or vaginal or conditions over.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DEFFIEUX, Principal Investigator — AP-HP, Antoine Béclère Hospital
Locations (1):
- Xavier DEFFIEUX, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided